CLINICAL TRIAL: NCT06030180
Title: CLUE: CLinical Utility Study of EsoGuard on Samples Collected Using EsoCheck as a Triage Test for Endoscopy to Identify Barrett's Esophagus (BE)
Brief Title: CLUE: CLinical Utility Study of EsoGuard
Acronym: PR-0410
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lucid Diagnostics, Inc. (Industry)
Responsible Party: Sponsor
Organization: PAVmed Inc. (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PR-0410
Record Dates: First submitted 2023-08-25; First posted 2023-09-08 (Actual); Last update posted 2025-06-27 (Actual); Status verified 2025-06

CONDITIONS: Barrett Esophagus; Barretts Esophagus With Dysplasia; Esophagus Adenocarcinoma
MeSH Terms: conditions — Barrett Esophagus; Adenocarcinoma Of Esophagus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Single Arm Study (Other)
  Interventions: Device: EsoGuard

INTERVENTIONS:
Device: EsoGuard — EsoGuard is a set of genetic assays and algorithms for the assessment of specific methylation patterns of DNA encoding the genes vimentin (VIM) and cyclin A1 (CCNA1)
  Other Names: EsoGuard test on cells collected using EsoCheck

SUMMARY:
Utilize real-world data from the commercial use of EsoGuard testing on samples collected with EsoCheck (EC/EG) to evaluate the impact of EsoGuard results on health care provider's decision for endoscopy referral. Assess patient compliance with recommendations for upper endoscopy, and relationship of compliance to positive EsoGuard results.

ELIGIBILITY:
Inclusion Criteria:

1. Individuals in whom the clinical decision has been made to screen for BE using EC/EG
2. Individuals who meet criteria for BE screening in accordance with either the 2022 ACG guidelines, or the AGA best practice advice from their 2022 clinical practice update.

Exclusion Criteria:

1. Individuals who fall outside the eligible population defined by the EsoCheck device Instructions For Use (IFU)
2. Individuals who do not meet either the ACG or AGA guidelines/practice advice for BE screening
3. Inability to provide written informed consent or participate in the required follow up

Ages: 12 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 566 (Actual)
Dates: Start 2023-02-23 (Actual); Primary Completion 2024-12-13 (Actual); Study Completion 2024-12-13 (Actual)

PRIMARY OUTCOMES:
Clinical Utility | Through study completion, an average of 1 year
  Utilize real-world data from the commercial use of EsoGuard testing on samples collected with EsoCheck (EC/EG) to evaluate the impact of EsoGuard results on health care provider's decision for endoscopy referral. This will be measured by asking physicians how the EsoGuard result impacted their referral decision.

SECONDARY OUTCOMES:
Patient Compliance | Through study completion, an average of 1 year
  Assess patient compliance with recommendations for upper endoscopy, and relationship of compliance to positive EsoGuard results. This will be measured by collecting data on whether patients received an endoscopy after being referred.

CONTACTS AND LOCATIONS:
Overall Officials: Gisella Lopez, Study Director — Lucid Diagnostics
Locations (8):
- United States (8):
  - Arkansas Heartburn Treatment Center, Heber Springs, Arkansas
  - Arvada West Family Medicine,, Arvada, Colorado
  - Colorado Primary Healthcare, Littleton, Colorado
  - Savii Health, Savannah, Georgia
  - James E Race, Dallas, Texas
  - Texas Digestive Specialists, Harlingen, Texas
  - Gastroenterology Partners of North Houston, PLLC, Shenandoah, Texas
  - Premier Family Medical, Lindon, Utah

IPD SHARING:
Plan to Share IPD: No